CLINICAL TRIAL: NCT04218318
Title: Safe Threshold to Discontinue Phototherapy in Term and Late Preterm Infant With Hemolytic Disease of Newborn: A Randomized Controlled Trial
Brief Title: Safe Threshold to Discontinue Phototherapy in Hemolytic Disease of Newborn
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Fatema Sulaiman Alhazmi, Cilinical fellow, Madinah Maternity and Children's Hospital, NICU, Ministry of Health, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-03-M-084
Record Dates: First submitted 2019-12-18; First posted 2020-01-06 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Hemolytic Disease of Newborn; Neonatal Hyperbilirubinemia
Keywords: Jaundice; Newborn; Hyperbilirubinemia; Rebound hyperbilirubinemia; Phototherapy; Hemolysis
MeSH Terms: conditions — Erythroblastosis, Fetal; Hyperbilirubinemia, Neonatal; Jaundice; Hyperbilirubinemia; Hemolysis | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: A prospective open labeled randomized control trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-threshold group (Active Comparator): Neonates in the low-threshold group phototherapy will be stopped if TSB reached ˃100 µmol/L below the AAP phototherapy threshold.
  Interventions: Device: phototherapy
- High-threshold group (Active Comparator): Neonates in high-threshold group phototherapy will be ceased if TSB level is 50-100 µmol/L below the appropriate AAP phototherapy threshold.
  Interventions: Device: phototherapy

INTERVENTIONS:
Device: phototherapy — Phototherapy will be commenced for neonates in both groups according to AAP guidelines.Neonates will be treated with intensified overhead blue LEDs phototherapy if they have a TSB level at or above phototherapy threshold. Neonates will be started on intensified 360◦ LED phototherapy if they have TSB level within 50µmol/L below the exchange threshold. The administration of IVIG is indicated in infants with isoimmune hemolytic disease if TSB lies within 34 to 51 micromol/L of the threshold for exchange transfusion and not responding to initial intensified phototherapy.Infants with a TSB concentration above the thresholds for exchange should have immediate intensified 360◦ LED phototherapy, and preparation for exchange transfusion will be started.Infants showed clinical signs of acute bilirubin encephalopathy will have an immediate exchange transfusion.

SUMMARY:
We hypothesized that adopting a lower rather than a higher threshold for phototherapy discontinuation will be associated with reduced rates of rebound hyperbilirubinemia in term and late preterm neonates with hemolytic disease of newborn.

Objectives: The investigators aimed to compare the safety of implementing low-threshold, compared to high- threshold, of TSB for phototherapy interruption in term and late preterm neonates with hemolytic disease of newborn.

DETAILED DESCRIPTION:
Neonates in high-threshold group phototherapy will be ceased if TSB level is 50-100 µmol/L below the appropriate 2004 AAP phototherapy threshold, whereas neonates in the low-threshold group phototherapy will be stopped if TSB reached ˃100 µmol/L below the AAP threshold.

Phototherapy will be commenced for neonates in both groups according to AAP guidelines.Neonates will be treated with intensified overhead blue LEDs phototherapy if they have a TSB level at or above phototherapy threshold. Neonates will be started on intensified 360◦ LED phototherapy if they have TSB level within 50µmol/L below the exchange threshold. The administration of IVIG is indicated in infants with isoimmune hemolytic disease if TSB lies within 34 to 51 micromol/L of the threshold for exchange transfusion and not responding to initial intensified phototherapy.Infants with a TSB concentration above the thresholds for exchange should have immediate intensified 360◦ LED phototherapy, and preparation for exchange transfusion will be started.Infants showed clinical signs of acute bilirubin encephalopathy will have an immediate exchange transfusion.

ELIGIBILITY:
Inclusion Criteria:

Healthy term and late-preterm neonates more than or equal 35 weeks gestation with hemolytic disease of newborn will be included. Enrolled infants should have evidence of hemolysis as defined by any of the following criteria:

1. positive DAT and blood group iso-immunization (ABO / RH incompatibility);and /or
2. HGB decline by 2g/dl within 24hour.

Exclusion Criteria:

* Major congenital abnormalities,
* Surgical problems,
* Direct hyperbilirubinemia
* Sepsis

Ages: 1 Hour to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Rebound hyperbilirubinemia | 28 days
  Number of participants of whome concentration of total serum bilirubin returned to or beyond the AAP phototherapy threshold within 72 hours of phototherapy discontinuation of a neonate's first round of phototherapy treatment.

SECONDARY OUTCOMES:
Duration of phototherapy | 28 days
  Duration of phototherapy
Length of hospital stay | 28 days
  Length of hospital stay
Adverse effects related to phototherapy | 28 days
  Number of participants who will develop erythematous rash, loose stool, hyperthermia, and dehydration
Rebound hyperbilirubinemia between 3-7 days after phototherapy stoppage | 28 days
  Number of participants of whome concentration of total serum bilirubin returned to or beyond the AAP phototherapy threshold between 3-7 days of phototherapy discontinuation of a neonate's first round of phototherapy treatment.
Rebound TSB level that exceeded the appropriate AAP phototherapy threshold by ≥35 µmol/L after phototherapy stoppage | 28 days
  Rebound TSB level that exceeded the appropriate AAP phototherapy threshold by ≥35 µmol/L after phototherapy stoppage
Rebound TSB level that exceeded the appropriate AAP exchange transfusion threshold after phototherapy storage | 28 days
  Number of participants of whome rebound TSB level that exceeded the appropriate AAP exchange transfusion threshold after phototherapy storage
Total Cost of NICU Care | 90 days
  Total Cost of NICU Care

CONTACTS AND LOCATIONS:
Overall Officials: Fatimah S Alhazmi, MD, Principal Investigator — Ministry of Health, Saudi Arabia
Locations (1):
- Madinah maternity and children's hospital, Madinah, Saudi Arabia